CLINICAL TRIAL: NCT06066177
Title: Impact of Triglyceride-Glucose Index on Cardiovascular Outcomes in Patients Presented With Myocardial Infarction With Nonobstructive Coronary Arteries
Brief Title: Impact of Triglyceride-Glucose Index on Cardiovascular Outcomes in Patients Presented With MINOCA
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Gamal Thabit Mohamed, Resident , department of Cardiology،Principal Investigator, Assiut University
Other Study IDs: TyG index and MINOCA
Record Dates: First submitted 2023-09-27; First posted 2023-10-04 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Major Cardiovascular Events
Keywords: Triglyceride glucose index Myocardial infarction MINOCA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Triglyceride glucose index TyG — Triglyceride glucose index is an indicator of insulin resistance

SUMMARY:
This work was designed to explore the role of the triglyceride-glucose (TyG) index in the prediction of cardiovascular outcomes in Patients Presented with myocardial infarction with nonobstructive coronary arteries.

DETAILED DESCRIPTION:
Acute myocardial infarction (AMI) remains the leading causes of high morbidity and mortality worldwide . Recently, a distinct population with myocardial infarction with nonobstructive coronary arteries (MINOCA) has been increasingly recognized because of the widespread use of coronary angiography. MINOCA occurs in 5%-10% of all AMI and they are younger and more often women compared to patients with AMI and obstructive coronary artery disease (CAD). The underlying causes of MINOCA are manifold and may include plaque rupture or erosion, thromboembolism, coronary spasm, spontaneous dissection, microvascular dysfunction and supply/demand mismatch. Some non-ischemic diseases such as myocarditis may also mimic the presentation of MINOCA . Of note, several studies have found that the prognosis of MINOCA is not trivial and patients are still at considerable risks for long-term adverse cardiovascular (CV) events despite the optimal secondary prevention treatments . Thus, it is of necessity and profound implications to find potential residual risk factors and improve prognosis in MINOCA population.

Insulin resistance (IR), a critical mechanism of the pathogenesis of diabetes, not only contributes to the development of cardiovascular diseases (CVD), but also significantly correlates with adverse CV outcomes. Additionally, IR often coexists with obesity, hypertension, and dyslipidemia , and all of these are well-known risk factors of CVD. Recently, the triglyceride-glucose (TyG) index derived from fasting triglyceride (TG) and fasting blood glucose (FBG) levels has been proposed as a new and valid surrogate indicator of IR . Till now, many studies have found that the TyG index is positively correlated with metabolic disorders, arterial stiffness , carotid atherogenesis , coronary artery calcification , and subclinical or symptomatic CAD. Moreover, growing evidence has showed that the TyG index is an independent predictor of poor CV outcomes in general population and in different cohorts with CAD, including patients with AMI or acute coronary syndrome (ACS) with or without diabetes

ELIGIBILITY:
Inclusion Criteria:

* All patients; diagnosed with myocardial infarction with nonobstructive coronary arteries (MINOCA)
* clinical symptoms
* ECG : ischemic changes with or without ST segment elevation
* Echocardiograpy : segmental wall motion abnormalities (SWMA)
* positive cardiac enzymes
* Coronary angiography: insignificant lesions ,the absence of culprit obstructive coronary artery disease (epicardial coronary artery stenosis ≥50%)

Exclusion Criteria:

* All non confirmed diagnosis of MINOCA
* cardiac

  * non-ischemic cardiomyopathies
* non-cardiac

  * pulmonary embolism
  * stroke
  * sepsis
  * ARDS

Max Age: 80 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Myocardial infarction patients who were underwent PPCI and the coronary angiography showing insignificant lesions (stenosis less than 50% )
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-01-20 (Estimated); Primary Completion 2028-08-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of major adverse cardiovascular events (MACE) | along one year follow up .
  including
  * all-cause death,
  * reinfarction,
  * stroke,
  * re-intervention
  * hospitalization for unstable angina or heart failure)

CONTACTS AND LOCATIONS:
Overall Officials: Ayman khairy Mohamed Hassan, Principal Investigator — Cardiology department; Khaled Mohamed Abdullah Mohamed, Principal Investigator — Cardiology department

REFERENCES:
- [Background] Gao S, Ma W, Huang S, Lin X, Yu M. Impact of triglyceride-glucose index on long-term cardiovascular outcomes in patients with myocardial infarction with nonobstructive coronary arteries. Nutr Metab Cardiovasc Dis. 2021 Oct 28;31(11):3184-3192. doi: 10.1016/j.numecd.2021.07.027. Epub 2021 Aug 4. PMID 34511291
- [Background] Zhao X, Wang Y, Chen R, Li J, Zhou J, Liu C, Zhou P, Sheng Z, Chen Y, Song L, Zhao H, Yan H. Triglyceride glucose index combined with plaque characteristics as a novel biomarker for cardiovascular outcomes after percutaneous coronary intervention in ST-elevated myocardial infarction patients: an intravascular optical coherence tomography study. Cardiovasc Diabetol. 2021 Jun 28;20(1):131. doi: 10.1186/s12933-021-01321-7. PMID 34183007